CLINICAL TRIAL: NCT06073119
Title: A Phase 2, International, Multicenter, Randomized, Double-blind, Placebo-controlled, Dose-ranging Study of Efficacy and Safety of SAR441566 in Adults With Moderate to Severe Plaque Psoriasis
Brief Title: A Study to Evaluate Efficacy and Safety of SAR441566 in Adults With Plaque Psoriasis
Acronym: SPECIFI-PSO
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: DRI17849; 2023-503911-14 (Registry Identifier: CTIS); U1111-1290-5787 (Registry Identifier: ICTRP); 2023-503911-14-00 (Registry Identifier: CTIS); 2023-503911-14 (EudraCT Number)
Record Dates: First submitted 2023-10-04; First posted 2023-10-10 (Actual); Results first posted 2025-11-10 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-10

CONDITIONS: Psoriasis
MeSH Terms: conditions — Psoriasis

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (6):
- SAR441566 dose regimen A (Experimental): Participants received dose regimen A of SAR441566
  Interventions: Drug: SAR441566
- SAR441566 dose regimen B (Experimental): Participants received dose regimen B of SAR441566
  Interventions: Drug: SAR441566
- SAR441566 dose regimen C (Experimental): Participants received dose regimen C of SAR441566
  Interventions: Drug: SAR441566
- SAR441566 dose regimen D (Experimental): Participants received dose regimen D of SAR441566
  Interventions: Drug: SAR441566
- SAR441566 dose regimen E (Experimental): Participants received dose regimen E of SAR441566
  Interventions: Drug: SAR441566
- Placebo (Placebo Comparator): Participants received SAR441566 matching placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SAR441566 — Tablet
  Arms: SAR441566 dose regimen A; SAR441566 dose regimen B; SAR441566 dose regimen C; SAR441566 dose regimen D; SAR441566 dose regimen E
Drug: Placebo — Tablet
  Arms: Placebo

SUMMARY:
This was a Phase 2, international, multicenter, randomized, double-blind, placebo-controlled, dose-ranging, 12-week study. It was designed to assess the therapeutic dose, efficacy, and safety of treatment with SAR441566 in male and female adults with moderate to severe plaque psoriasis. Study details included a screening period (4 weeks and not less than 11 days before Day 1), a treatment period (12 weeks ± 3 days) and a post-treatment period (safety follow-up) (4 weeks ± 3 days). The total number of study visits was 7.

DETAILED DESCRIPTION:
The overall study duration for each participant was up to 149 days.

ELIGIBILITY:
Inclusion Criteria:

* Participants with moderate to severe plaque psoriasis for at least 6 months, meeting the following criteria at screening and D1 (prior to randomization):

  * PASI ≥ 12 points;
  * and sPGA score ≥ 3 points;
  * and BSA score ≥ 10%
* Had to be a candidate for phototherapy or systemic therapy.
* Total body weight ≥ 50 kg (110 lb) and body mass index (BMI) within the range [18 - 35] kg/m^2 (inclusive)

Exclusion Criteria:

* Other forms of psoriasis than plaque psoriasis, such as guttate psoriasis, psoriatic arthritis, or pustular psoriasis. Nail psoriasis was accepted for inclusion.
* Plaque psoriasis was restricted to scalp, palms, soles, or flexures only.
* Any other skin diseases that could interfere with psoriasis evaluation or treatment response (eg, atopic dermatitis, fungal or bacterial superinfection)
* Other immunologic (autoimmune or inflammatory) disorder, except medically controlled diabetes or thyroid disorder as per Investigator's judgement
* History of recurrent or recent serious infection (eg, pneumonia, septicemia), or infection(s) requiring hospitalization or treatment with IV antiinfectives (antibiotics, antivirals, antifungals, antihelminthics) within 30 days prior to D1, or infections(s) requiring oral antiinfectives (antibiotics, antivirals, antifungals, antihelminthics) within 14 days prior to D1
* Known history of or suspected significant current immunosuppression, including history of invasive opportunistic or helminthic infections despite infection resolution or otherwise recurrent infections of abnormal frequency or prolonged duration
* Participant with personal or family history of long QT syndrome
* History of moderate to severe congestive heart failure (New York Heart Association Class III or IV), or recent cerebrovascular accident, or any other condition in the opinion of the Investigator that would have put the participant at risk by participation in the protocol
* History of solid organ transplant
* History of alcohol or drug abuse within the past 2 years
* History of diagnosis of demyelinating disease such as but not limited to:

  * Multiple Sclerosis
  * Acute Disseminated Encephalomyelitis
  * Balo's Disease (Concentric Sclerosis)
  * Charcot-Marie-Tooth Disease
  * Guillain-Barre Syndrome
  * Human T-lymphotropic virus 1 Associated Myelopathy
  * Neuromyelitis Optica (Devic's Disease)
* Planned surgery during the treatment period
* Active malignancy, lymphoproliferative disease, or malignancy in remission for less than 5 years, except adequately treated (cured) localized carcinoma in situ of the cervix or ductal breast, or squamous cell carcinoma, or basal cell carcinoma of the skin
* Any live (attenuated) vaccine within 6 weeks prior to randomization (eg, varicella zoster vaccine, oral polio, rabies) or planned to receive one during the trial

The above information was not intended to contain all considerations relevant to a potential participation in a clinical trial

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 221 (Actual)
Dates: Start 2023-10-26 (Actual); Primary Completion 2024-11-13 (Actual); Study Completion 2024-12-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences and Operations, Study Director — Sanofi
Locations (51):
- United States (11):
  - Scottsdale Clinical Trials Site Number : 8400025, Scottsdale, Arizona
  - Dermatology Research Associates- Site Number : 8400019, Los Angeles, California
  - Daxia Trials Site Number : 8400022, Boca Raton, Florida
  - Renaissance Research and Medical Group, Inc- Site Number : 8400018, Cape Coral, Florida
  - Driven Research, LLC- Site Number : 8400012, Coral Gables, Florida
  - FXM Clinical Research Ft. Lauderdale, LLC Site Number : 8400015, Fort Lauderdale, Florida
  - Direct Helpers Medical Center Inc- Site Number : 8400023, Hialeah, Florida
  - FXM Clinical Research Miami, LLC- Site Number : 8400016, Miami, Florida
  - Center for Clinical Studies, LTD. LLP- Site Number : 8400007, Houston, Texas
  - Center for Clinical Studies, LTD, LLP- Site Number : 8400013, Webster, Texas
  - Jordan Valley Dermatology Center- Site Number : 8400027, South Jordan, Utah
- Argentina (3):
  - Investigational Site Number : 0320003, CABA, Buenos Aires
  - Investigational Site Number : 0320001, Buenos Aires, Buenos Aires F.D.
  - Investigational Site Number : 0320002, CABA, Buenos Aires F.D.
- Investigational Site Number : 1000001, Sofia, Bulgaria
- Canada (2):
  - Investigational Site Number : 1240006, London, Ontario
  - Investigational Site Number : 1240002, Waterloo, Ontario
- Chile (4):
  - Investigational Site Number : 1520003, Santiago, Reg Metropolitana de Santiago
  - Investigational Site Number : 1520001, Santiago, Reg Metropolitana de Santiago
  - Investigational Site Number : 1520004, Santiago, Reg Metropolitana de Santiago
  - Investigational Site Number : 1520002, Santiago, Reg Metropolitana de Santiago
- China (2):
  - Investigational Site Number : 1560001, Hangzhou
  - Investigational Site Number : 1560002, Wuxi
- Investigational Site Number : 2030003, Brno, Czechia
- Georgia (2):
  - Investigational Site Number : 2680002, Batumi
  - Investigational Site Number : 2680001, Tbilisi
- Germany (3):
  - Investigational Site Number : 2760004, Blankenfelde-Mahlow
  - Investigational Site Number : 2760001, Frankfurt am Main
  - Investigational Site Number : 2760002, Witten
- Hungary (2):
  - Investigational Site Number : 3480003, Budapest
  - Investigational Site Number : 3480002, Debrecen
- Japan (6):
  - Investigational Site Number : 3920004, Kamimashiki Gun, Kumamoto
  - Investigational Site Number : 3920003, Sakai-shi, Osaka
  - Investigational Site Number : 3920006, Itabashi-ku, Tokyo
  - Investigational Site Number : 3920002, Tachikawa-shi, Tokyo
  - Investigational Site Number : 3920005, Ichikawa-shi
  - Investigational Site Number : 3920001, Yokohama
- Investigational Site Number : 4800001, Quatre Bornes, Mauritius
- Poland (2):
  - Investigational Site Number : 6160001, Bydgoszcz
  - Investigational Site Number : 6160002, Katowice
- Portugal (3):
  - Investigational Site Number : 6200003, Guimarães
  - Investigational Site Number : 6200002, Lisbon
  - Investigational Site Number : 6200001, Lisbon
- Spain (5):
  - Investigational Site Number : 7240003, Manises, Valencia
  - Investigational Site Number : 7240007, Alicante
  - Investigational Site Number : 7240005, Madrid
  - Investigational Site Number : 7240004, Madrid
  - Investigational Site Number : 7240002, Zaragoza
- Turkey (Türkiye) (2):
  - Investigational Site Number : 7920002, Antalya
  - Investigational Site Number : 7920001, Kayseri
- Investigational Site Number : 8260001, Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized, and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- See also: DRI17849 Plain Language Results Summary — https://sanofi.trialsummaries.com/Study/StudyDetails?id=25536&tenant=MT_SNY_9011

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 51 centers in 17 countries. A total of 292 participants were screened from 26 October 2023 to 24 July 2024, of which 71 were screen failures. Screen failures were mainly due to not meeting the eligibility criteria.
Pre-assignment Details: 221 participants were randomized in 2 different strata: naïve targeted immunotherapy population (NTIP) and experienced targeted immunotherapy population (ETIP). 147 participants were randomized into NTIP in 1:1:1:1:1:1 ratio to receive either placebo or SAR441566 at 200 mg BID, 100 mg BID, 200 mg QD, 100 mg QD or 50 mg QD. 74 participants were randomized into ETIP in 2:2:2:1 ratio to receive either placebo or SAR441566 at 200 mg BID, 200 mg QD, 100 mg QD. ETIP was used for exploratory analysis.
Groups:
- Placebo: Participants received placebo matched to SAR441566 orally from Day 1 up to 12 weeks.
- SAR441566 200 mg BID: Participants received 200 milligrams (mg) twice a day (BID) of SAR441566 orally from Day 1 up to 12 weeks.
- SAR441566 100 mg BID: Participants received 100 mg BID of SAR441566 orally from Day 1 up to 12 weeks.
- SAR441566 200 mg QD: Participants received 200 mg once a day (QD) of SAR441566 orally from Day 1 up to 12 weeks.
- SAR441566 100 mg QD: Participants received 100 mg QD of SAR441566 orally from Day 1 up to 12 weeks.
- SAR441566 50 mg QD: Participants received 50 mg QD of SAR441566 orally from Day 1 up to 12 weeks.
Period: Overall Study
Arm/Group | Placebo | SAR441566 200 mg BID | SAR441566 100 mg BID | SAR441566 200 mg QD | SAR441566 100 mg QD | SAR441566 50 mg QD
Started | 35 | 47 | 24 | 46 | 45 | 24
Completed | 27 | 36 | 20 | 41 | 39 | 23
Not Completed | 8 | 11 | 4 | 5 | 6 | 1
Not completed — Adverse Event | 1 | 3 | 0 | 0 | 1 | 0
Not completed — Non-compliance with study schedule | 1 | 0 | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 4 | 4 | 3 | 5 | 3 | 1
Not completed — Other | 2 | 4 | 1 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: The randomized population included all participants from screened population who were allocated to a randomized study treatment by interactive web response system regardless of whether the study treatment was received.
Groups:
- SAR441566 200 mg BID: Participants received 200 mg BID of SAR441566 orally from Day 1 up to 12 weeks.
- SAR441566 200 mg QD: Participants received 200 mg QD of SAR441566 orally from Day 1 up to 12 weeks.
- Total: Total of all reporting groups
Arm/Group | Placebo | SAR441566 200 mg BID | SAR441566 100 mg BID | SAR441566 200 mg QD | SAR441566 100 mg QD | SAR441566 50 mg QD | Total
Number analyzed (Participants) | 35 | 47 | 24 | 46 | 45 | 24 | 221
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.0 (13.0) | 43.5 (13.7) | 45.5 (11.0) | 45.4 (13.9) | 46.8 (12.9) | 38.4 (13.2) | 44.3 (13.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 14 | 10 | 12 | 13 | 13 | 75
  Male | 22 | 33 | 14 | 34 | 32 | 11 | 146
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 5 | 7 | 6 | 8 | 4 | 2 | 32
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 1 | 2 | 0 | 3
  Black or African American | 0 | 1 | 2 | 0 | 2 | 1 | 6
  White | 29 | 38 | 14 | 37 | 37 | 21 | 176
  More than one race | 0 | 0 | 1 | 0 | 0 | 0 | 1
  Unknown or Not Reported | 1 | 1 | 1 | 0 | 0 | 0 | 3

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With a 75% or Greater Psoriasis Area and Severity Index (PASI) Score Reduction From Baseline (PASI75) at Week 12
Description: PASI is linear combination of percent of surface area of skin that is affected and severity of erythema(E),induration(i),desquamation(D) over 4 body regions: head(h),trunk(t),upper extremities(u),lower extremities(l). The signs of severity, E, i and D of lesions are assessed using numeric scale for which scores are made independently for each of the areas; range:0 (complete lack of cutaneous involvement) to 4 (severest possible involvement). For each body area, percentage of considered body area covered by plaque psoriasis is translated into numerical value "Ax":0=no involvement,1=<10% to 6=90 to 100% involvement. These scores are noted Ah, At, Au, and Al in formula below. The PASI score is calculated according to the following formula: PASI = 0.1(Eh+ih+Dh)Ah + 0.3(Et+it+Dt)At + 0.2(Eu+iu+Du)Au + 0.4(El+il+Dl)Al. PASI score range:0 (no disease) to 72 (maximal disease);higher scores: greater psoriasis severity. Percentage of participants with PASI75 at Week 12 is presented.
Time Frame: Baseline (Day 1) and Week 12
Population: The NTIP included all randomized participants who never received targeted immunotherapy for psoriasis.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | SAR441566 200 mg BID | SAR441566 100 mg BID | SAR441566 200 mg QD | SAR441566 100 mg QD | SAR441566 50 mg QD
Number analyzed (Participants) | 25 | 25 | 24 | 24 | 25 | 24
percentage of participants | 20.0 | 44.0 | 50.0 | 58.3 | 28.0 | 33.3
Statistical Analysis 1: Comparison: Placebo vs SAR441566 200 mg BID; Test type: Superiority; p = 0.0874, Cochran-Mantel-Haenszel — A hierarchical testing was used to control the overall type I error of 0.05 (two-sided). Testing was performed in the order of 200 mg BID, 100 mg BID, 200 mg QD versus placebo; Adjusted for baseline PASI score (<=20, >20); Response rate difference (RRD), % = 23.43, 95% CI 2-sided [-2.74 to 45.98] — Difference = SAR441566 Dose Regimen 200 mg BID - placebo
Statistical Analysis 2: Comparison: Placebo vs SAR441566 100 mg BID; Test type: Superiority; p = 0.0185, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; Adjusted for baseline PASI score (<=20, >20); RRD, % = 33.08, 95% CI 2-sided [5.71 to 54.83] — Difference = SAR441566 Dose Regimen 100 mg BID - placebo
Statistical Analysis 3: Comparison: Placebo vs SAR441566 200 mg QD; Test type: Superiority; p = 0.0077, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; Adjusted for baseline PASI score (<=20, >20); RRD, % = 38.02, 95% CI 2-sided [10.62 to 58.84] — Difference = SAR441566 Dose Regimen 200 mg QD - placebo
Statistical Analysis 4: Comparison: Placebo vs SAR441566 100 mg QD; Test type: Superiority; p = 0.4576, Cochran-Mantel-Haenszel — No multiplicity adjustment, hence p-value is nominal; Adjusted for baseline PASI score (<=20, >20); RRD, % = 9.35, 95% CI 2-sided [-14.72 to 32.40] — Difference = SAR441566 Dose Regimen 100 mg QD - placebo
Statistical Analysis 5: Comparison: Placebo vs SAR441566 50 mg QD; Test type: Superiority; p = 0.3051, Cochran-Mantel-Haenszel — No multiplicity adjustment, hence p-value is nominal; Adjusted for baseline PASI score (<=20, >20); RRD, % = 13.44, 95% CI 2-sided [-11.38 to 36.72] — Difference = SAR441566 Dose Regimen 50 mg QD - placebo

2. Secondary Outcome: Percent Change From Baseline in Psoriasis Area and Severity Index to Week 12
Description: PASI is linear combination of percent of surface area of skin that is affected and severity of E, i, D over 4 body regions: h, t, u, l. The signs of severity, E, i and D of lesions are assessed using numeric scale for which scores are made independently for each of the areas; range: 0 (complete lack of cutaneous involvement) to 4 (severest possible involvement). For each body area, percentage of considered body area covered by plaque psoriasis is translated into numerical value "Ax": 0= no involvement,1= <10% to 6 =90 to 100% involvement. These scores are noted Ah, At, Au, and Al in formula below. The PASI score is calculated according to the following formula: PASI = 0.1(Eh+ih+Dh)Ah + 0.3(Et+it+Dt)At + 0.2(Eu+iu+Du)Au + 0.4(El+il+Dl)Al. The PASI score ranges from 0 (no disease) to 72 (maximal disease); higher scores indicate greater psoriasis severity. Baseline was defined as last available value before the first dose of study treatment.
Time Frame: Baseline (Day 1) to Week 12
Population: The NTIP included all randomized participants who never received targeted immunotherapy for psoriasis.
Measure: Least Squares Mean (95% Confidence Interval); unit: percent change
Arm/Group | Placebo | SAR441566 200 mg BID | SAR441566 100 mg BID | SAR441566 200 mg QD | SAR441566 100 mg QD | SAR441566 50 mg QD
Number analyzed (Participants) | 25 | 25 | 24 | 24 | 25 | 24
percent change | -40.65 [-52.98 to -28.33] | -63.42 [-75.73 to -51.11] | -60.56 [-73.12 to -48.01] | -65.18 [-77.74 to -52.62] | -60.84 [-73.14 to -48.54] | -65.85 [-78.40 to -53.30]

3. Secondary Outcome: Percentage of Participants With Static Psoriasis Global Assessment (sPGA) Score 0 (Complete Clearance) or 1 (Minimal Disease) at Week 12
Description: sPGA is 5-point score based on average thickness,erythema,and scaling of all psoriatic lesions.Score ranges:E:0(normal) to 4(bright to deep red coloration of lesions); i (plaque elevation):0(none) to 4(severe thickening with hard edges; D:0(no scaling) to 3(moderate scaling).Overall scoring: average of E,i,D;range:0(clear)= 0 for all 3 symptoms; 1(almost clear)=mean >0, <1.5, normal to pink coloration, just detectable(possible slight elevation),no to minimal focal scaling; 2(mild)= mean >= 1.5, <2.5, pink to light red coloration, mild thickening, predominantly fine scaling; 3(moderate)= mean >=2.5,<3.5, dull to bright red coloration, clearly distinguishable to moderate thickening, moderate scaling; 4(severe)= mean >=3.5,bright to deep dark red coloration,severe thickening with hard edges,severe coarse scaling covering almost all or all lesions.Lower score:less body coverage,with 0:complete clearance and 1:minimal disease. Total participants who received score of 0 and 1 are reported.
Time Frame: Baseline (Day 1) and Week 12
Population: The NTIP included all randomized participants who never received targeted immunotherapy for psoriasis.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | SAR441566 200 mg BID | SAR441566 100 mg BID | SAR441566 200 mg QD | SAR441566 100 mg QD | SAR441566 50 mg QD
Number analyzed (Participants) | 25 | 25 | 24 | 24 | 25 | 24
percentage of participants | 24.0 | 36.0 | 54.2 | 58.3 | 36.0 | 50.0

4. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs), Treatment-Emergent Serious Adverse Events (TESAEs), Treatment-Emergent Adverse Events of Special Interest (TEAESIs), Study Treatment Discontinuation and Study Withdrawals Due to TEAEs
Description: An AE was any untoward medical occurrence in a clinical study participant, temporally associated with the use of study treatment, whether considered related to the study treatment. An SAE was defined as any untoward medical occurrence that, at any dose, resulted in death, was life-threatening, required inpatient hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability/incapacity, was a congenital anomaly/birth defect or was an important medical event. TEAEs were AEs that developed, worsened or became serious during the TE period. An AESI was an AE (serious or non-serious) of scientific and medical concern specific to the Sponsor's product or program, for which ongoing monitoring and immediate notification by the Investigator to the Sponsor was required.
Time Frame: From first dose of study treatment (Day 1) up to 5 days post last dose of study treatment, up to 102 days
Population: The safety population included all randomized participants who took at least 1 dose of study treatment, regardless of the amount of treatment administered.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | SAR441566 200 mg BID | SAR441566 100 mg BID | SAR441566 200 mg QD | SAR441566 100 mg QD | SAR441566 50 mg QD
Number analyzed (Participants) | 35 | 47 | 24 | 46 | 45 | 24
Participants
  Any TEAE | 12 | 27 | 9 | 26 | 7 | 8
  Any TESAE | 1 | 1 | 0 | 0 | 1 | 0
  Any TEAESI | 1 | 4 | 0 | 1 | 0 | 0
  Any TEAE leading to study treatment discontinuation | 1 | 5 | 0 | 1 | 1 | 0
  Any TEAE leading to study treatment withdrawal | 0 | 1 | 0 | 2 | 0 | 0

5. Secondary Outcome: Pre-Dose Plasma Concentration of SAR441566
Description: Blood samples were collected at indicated timepoints for the assessment of pre-dose plasma concentration of SAR441566.
Time Frame: 1 hour pre-dose on Weeks 2, 4, 8 and 12
Population: The pharmacokinetic (PK) population included all participants from the safety population with at least 1 post-baseline PK result with adequate documentation of dosing and sampling dates and times. Only those participants with data collected at specified timepoints are reported.
Measure: Mean (Standard Deviation); unit: nanogram per milliliter (ng/mL)
Arm/Group | SAR441566 200 mg BID | SAR441566 100 mg BID | SAR441566 200 mg QD | SAR441566 100 mg QD | SAR441566 50 mg QD
Number analyzed (Participants) | 39 | 20 | 38 | 38 | 23
nanogram per milliliter (ng/mL)
  Week 2: number analyzed (Participants) | 38 | 20 | 38 | 38 | 23
  Week 2 | 289.714 (178.652) | 115.745 (79.341) | 71.126 (33.287) | 32.581 (18.090) | 16.685 (9.880)
  Week 4: number analyzed (Participants) | 39 | 18 | 37 | 37 | 22
  Week 4 | 294.928 (193.309) | 110.083 (72.664) | 74.071 (41.391) | 31.011 (18.041) | 17.089 (10.061)
  Week 8: number analyzed (Participants) | 31 | 19 | 34 | 30 | 23
  Week 8 | 285.981 (200.600) | 101.216 (63.100) | 66.287 (50.241) | 34.729 (21.556) | 14.566 (14.117)
  Week 12: number analyzed (Participants) | 32 | 18 | 35 | 35 | 23
  Week 12 | 242.188 (151.416) | 86.317 (53.575) | 56.216 (34.269) | 30.711 (22.277) | 14.650 (10.029)

6. Secondary Outcome: Post-Dose Plasma Concentration of SAR441566
Description: Blood samples were collected at indicated timepoints for the assessment of post-dose plasma concentration of SAR441566.
Time Frame: 2.5 to 3.5 hours post-dose on Day 1, Weeks 2, 4, 8 and 12
Population: The PK population included all participants from the safety population with at least 1 post-baseline PK result with adequate documentation of dosing and sampling dates and times. Only those participants with data collected at specified timepoints are reported.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | SAR441566 200 mg BID | SAR441566 100 mg BID | SAR441566 200 mg QD | SAR441566 100 mg QD | SAR441566 50 mg QD
Number analyzed (Participants) | 46 | 22 | 42 | 43 | 24
ng/mL
  Day 1 | 135.396 (77.175) | 58.449 (25.096) | 132.462 (71.387) | 59.010 (34.099) | 33.008 (16.583)
  Week 2: number analyzed (Participants) | 12 | 12 | 8 | 12 | 9
  Week 2 | 438.750 (243.198) | 151.108 (72.612) | 158.463 (88.156) | 115.275 (49.937) | 56.667 (16.388)
  Week 4: number analyzed (Participants) | 40 | 21 | 39 | 40 | 22
  Week 4 | 432.998 (224.552) | 176.800 (87.429) | 184.854 (91.237) | 89.428 (45.908) | 45.145 (28.222)
  Week 8: number analyzed (Participants) | 9 | 10 | 4 | 10 | 8
  Week 8 | 428.111 (291.601) | 183.570 (101.811) | 222.750 (168.237) | 100.190 (59.421) | 51.175 (35.799)
  Week 12: number analyzed (Participants) | 33 | 20 | 34 | 36 | 22
  Week 12 | 401.897 (191.133) | 150.990 (80.672) | 153.229 (86.896) | 86.200 (41.862) | 42.877 (24.508)

ADVERSE EVENTS:
Time Frame: Adverse events were collected from first dose of study treatment (Day 1) up to 5 days post last dose of study treatment, up to 102 days. All-cause mortality (deaths) were collected from screening (Week -4) up to end of follow-up, 412 days.
Description: Analysis was performed on the safety population.
Arm/Group | Placebo | SAR441566 200 mg BID | SAR441566 100 mg BID | SAR441566 200 mg QD | SAR441566 100 mg QD | SAR441566 50 mg QD
All-Cause Mortality (participants affected / at risk) | 0/35 | 0/47 | 0/24 | 0/46 | 0/45 | 0/24
Serious Adverse Events (participants affected / at risk) | 1/35 | 1/47 | 0/24 | 0/46 | 1/45 | 0/24
Other Adverse Events (participants affected / at risk) | 12/35 | 27/47 | 9/24 | 26/46 | 6/45 | 8/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=35) | SAR441566 200 mg BID (N=47) | SAR441566 100 mg BID (N=24) | SAR441566 200 mg QD (N=46) | SAR441566 100 mg QD (N=45) | SAR441566 50 mg QD (N=24)
Staphylococcal Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Benign Pancreatic Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fracture Of Penis (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=35) | SAR441566 200 mg BID (N=47) | SAR441566 100 mg BID (N=24) | SAR441566 200 mg QD (N=46) | SAR441566 100 mg QD (N=45) | SAR441566 50 mg QD (N=24)
Nasopharyngitis (Infections and infestations) | 0 (0) | 5 (5) | 2 (2) | 2 (2) | 1 (1) | 3 (3)
Dysgeusia (Nervous system disorders) | 0 (0) | 5 (6) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 2 (2) | 2 (3) | 1 (2) | 3 (3) | 0 (0) | 1 (1)
Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Alanine Aminotransferase Increased (Investigations) | 2 (2) | 3 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood Alkaline Phosphatase Increased (Investigations) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abscess Limb (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Furuncle (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Gastroenteritis Viral (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Localised Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Upper Respiratory Tract Infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Viral Labyrinthitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Viral Upper Respiratory Tract Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Basal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Seborrhoeic Keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Idiopathic Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Decreased Appetite (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diabetic Metabolic Decompensation (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Irritability (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Post-Traumatic Stress Disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tension (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Burning Sensation (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eye Irritation (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Myocardial Infarction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Productive Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rhinitis Allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Abdominal Discomfort (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal Pain Upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dry Mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Faeces Soft (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Food Poisoning (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 2 (3) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatic Steatosis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Alopecia Areata (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dandruff (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Psoriasis (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Seborrhoeic Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Back Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rotator Cuff Syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal Pain (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Influenza Like Illness (General disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Malaise (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aspartate Aminotransferase Increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bilirubin Conjugated Increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood Bilirubin Increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood Creatine Phosphokinase Increased (Investigations) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Blood Creatinine Increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Electrocardiogram Qt Interval Abnormal (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hepatic Enzyme Increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neutrophil Count Decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
White Blood Cell Count Decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Accidental Overdose (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Foot Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Road Traffic Accident (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skin Abrasion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pregnancy Of Partner (Social circumstances) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor supports publication of clinical trial results but may request that investigators temporarily delay or alter publications in order to protect proprietary information. The Sponsor may also require that the results of multicenter studies be published only in their entirety and not as individual site data.

DOCUMENTS (2):
  • Study Protocol (2024-04-25): https://cdn.clinicaltrials.gov/large-docs/19/NCT06073119/Prot_000.pdf
  • Statistical Analysis Plan (2024-12-05): https://cdn.clinicaltrials.gov/large-docs/19/NCT06073119/SAP_001.pdf